CLINICAL TRIAL: NCT01199874
Title: The Immunogenicity of Rotavirus Vaccine Under Different Age Schedules and the Impact of Withholding Breast Feeding Around the Time of Vaccination on the Immunogenicity of Rotarix Vaccine
Brief Title: Immunogenicity of Rotavirus Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PATH HS534
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Rotavirus; Rotavirus vaccine; Dosing schedule; Immunogenicity; Breast feeding; Pakistan
MeSH Terms: conditions — Breast Feeding | interventions — Rotavirus Vaccines; RIX4414 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Primary 1: Rotavirus vaccine 6 and 10 weeks (Active Comparator): EPI vaccines + rotavirus vaccine at 6 and 10 weeks
  Interventions: Biological: Rotavirus vaccine
- Primary 1: Rotavirus vaccine 6, 10 and 14 weeks (Experimental): EPI vaccines + rotavirus vaccine at 6, 10 and 14 weeks
  Interventions: Biological: Rotavirus vaccine
- Primary 1: Rotavirus vaccine 10 and 14 weeks (Experimental): EPI vaccines + rotavirus vaccine at 10 and 14 weeks
  Interventions: Biological: Rotavirus vaccine
- Primary 2: Rotavirus vaccine withholding breast feeding (Experimental): EPI vaccines + rotavirus vaccine at 6, 10 and 14 weeks withholding breastfeeding
  Interventions: Biological: Rotavirus vaccine
- Primary 2: Rotavirus vaccine with immediate breast feeding (Experimental): EPI vaccines + rotavirus vaccine at 6, 10 and 14 weeks with immediate breastfeeding
  Interventions: Biological: Rotavirus vaccine
- Baseline seroconversion for rotavirus (No Intervention): EPI vaccines

INTERVENTIONS:
Biological: Rotavirus vaccine — live attenuated oral rotavirus vaccine; lyophilized; 1 ml
  Other Names: Rotarix
  Arms: Primary 1: Rotavirus vaccine 10 and 14 weeks; Primary 1: Rotavirus vaccine 6 and 10 weeks; Primary 1: Rotavirus vaccine 6, 10 and 14 weeks; Primary 2: Rotavirus vaccine with immediate breast feeding; Primary 2: Rotavirus vaccine withholding breast feeding

SUMMARY:
Rotavirus is one of the most common causes of severe diarrhea, responsible for 40% of all diarrhea related deaths in children worldwide. Two vaccines against Rotavirus, Rotarix® and Rotateq® were licensed in many high and middle income countries in 2006, but lack of efficacy data in low income countries had prevented WHO from making a universal recommendation of their use until recently. This study will be conducted in Pakistan and will look at two objectives:

1. To compare the immunogenicity of Rotarix® vaccine when administered at 6 and 10 weeks of life and at 6, 10 and 14 weeks of life.
2. To compare the immunogenicity of Rotarix® vaccine in infants breast fed at the time of vaccine administration with infants whose breast feeding is withheld for one hour before and after vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks 0 days to 6 weeks 6 days age at the time of enrollment.
* Healthy infant free of chronic or serious medical condition as determined by history and physical exam at time of enrollment into in the study.
* Written informed consent obtained from the parents or guardians.

Exclusion Criteria:

* Hypersensitivity to any of the vaccine components.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days of first dose of study vaccine or during the study.
* Use of any immunosuppressive drugs.
* Previous intussusception or abdominal surgery.
* Enrolment in any other trial (Simplified Antibiotic Therapy for Neonatal Sepsis Trial, Management of Omphalitis Trial).
* Birth weight less than 1500 grams; or if birth weight is unknown, weight less than 2000 grams on or before 28 days.
* Immunoglobulin and/or blood products use since birth or during the study period.

Ages: 6 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1140 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Seropositivity as anti-rotavirus IgA concentration >/= 20 U/ml | 6, 10, 14 and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S. Asad Ali, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Derived] Ali A, Kazi AM, Cortese MM, Fleming JA, Moon S, Parashar UD, Jiang B, McNeal MM, Steele D, Bhutta Z, Zaidi AK. Impact of withholding breastfeeding at the time of vaccination on the immunogenicity of oral rotavirus vaccine--a randomized trial. PLoS One. 2015 Jun 2;10(6):e0127622. doi: 10.1371/journal.pone.0127622. eCollection 2015. PMID 26035743